CLINICAL TRIAL: NCT03299621
Title: Anesthetic Depth Using PLE (Phase Lag Entropy)
Brief Title: Monitoring of Anesthetic Depth and EEG Band Power Using PLE (Phase Lag Entropy) During Propofol Anesthesia
Acronym: PLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Hye-Won Shin, Department of Anesthesiology and Pain Medicine, Korea University Anam Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: MD17014
Record Dates: First submitted 2017-08-25; First posted 2017-10-03 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLE (Phase Lag Entropy) monitoring (Experimental): Investigators monitor the change of PLE value using the sensor of PLEM™ during propofol anesthesia.
  Interventions: Device: PLE (Phase Lag Entropy)
- Muscle relaxant injection (Experimental): Investigators monitor the change for PLE value using the sensor of PLEM™ before and after the injection of muscle relaxant.
  Interventions: Drug: Muscle Relaxant

INTERVENTIONS:
Device: PLE (Phase Lag Entropy) — Monitoring of PLE value using the monitoring of PLEM™ device during propofol anesthesia.
  Other Names: PLEM™ (Inbody co., ltd)
  Arms: PLE (Phase Lag Entropy) monitoring
Drug: Muscle Relaxant — Monitoring of PLE value using the monitoring of PLEM™ device before and after the injection of muscle relaxant that used for tracheal intubation.
  Other Names: Muscle relaxant (rocuronium)
  Arms: Muscle relaxant injection

SUMMARY:
The evaluation of the anesthetic depth monitoring using PLE (Phase Lag Entropy) during propofol anesthesia

DETAILED DESCRIPTION:
The devices using EEG are commonly used for measuring the depth of consciousness during anesthesia. However, the existing devices are largely dependent on the biphasic analysis of 1-channel EEG signals, and thus do not provide proper information for anesthetic depth.

Recent study reported that the complexity or diversity of communication between the brain regions is related to the level of consciousness. In particular, during anesthesia, the phase synchronization (phase shift) between EEG signals at the front of the brain increases, indicating a reduction in communication diversity and a close relationship with loss of consciousness. Therefore, to predict the depth of sleep, a technique for precisely quantifying the complexity of inter-domain communication in the frontal brain is needed. Recently, PLEM™ (Inbody co., ltd, Republic of Korea), developed using the phase lag entropy (PLE), is a 4-channel EEG monitoring device that measures the entropy of the phase difference pattern between two channels of prefrontal and frontal brain. In addition, PLEM™ is able to observe changes in band power of EEG (Gamma, Beta, Alpha, Theta, and Delta waves). As the depth of anesthesia increases, the amplitude and frequency of EEG decreases. Generally, Beta waves (13-30 Hz) are seen in awake conscious patients and Alpha waves (8-12 Hz) are seen in patients resting with eyes closed. And Theta waves (4-7 Hz) and Delta waves (0-3 Hz) can be present in a patient who is sleeping or anesthetized.

The purpose of this study was to evaluate the efficacy for anesthetic depth monitoring of PLEM™ monitor during propofol anesthesia. The primary outcome of this study was to investigate the changes of PLE value and band power of EEG (Gamma, Beta, Alpha, Theta, Delta waves) on the PLEM™ monitor while varying the depth of anesthesia using propofol target controlled infusion (TCI) during anesthetic induction. The secondary outcomes of this study were to investigate whether the muscle relaxant affects the PLE value, and to compare the PLE values with BIS (bispectral index) (Aspect medical system, USA) that was the most widely used to measure the depth of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* The patients undergoing elective general anesthesia with American Society fo Anesthesiologist (ASA) physical status I or II (20-60 years)

Exclusion Criteria:

* Patients with difficulty airway
* Patients with cardiovascular disease
* Patients with cerebrovascular disease
* Patients with respiratory disease

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
PLE (Phase Lag Entropy) value before and after intubation | at the time points that propofol target effect site concentration reach to 0, 2, 4, 5, 6 μg/ml, and the time points before and after intubation
  Investigators measure the PLE value at the time points that propofol target effect site concentration reach at 0, 2, 4, 5, 6 μg/ml, and the time points before and after intubation.

SECONDARY OUTCOMES:
PLE value before and after the injection of muscle relaxant | at 3 min after the injection of muscle relaxant, immediately after intubation
  Investigators measure the PLE value before the injection of muscle relaxant, at 3 min after the injection of muscle relaxant, and immediately after intubation.
PLE value and BIS value at that time of induction and awakening | at the time point of no-response to verbal command during induction (modified Observer's assessment of Alertness/Sedation scale (modified OAA/S scale) = 2, at the time point of response to verbal command during awakening (modified OAA/S scale = 3).
  Investigators measure the PLE value and BIS value at the time point of no-response to verbal command during induction ('modified Observer's assessment of Alertness/Sedation scale (modified OAA/S scale) = 2], at the time point of response to verbal command during awakening [modified OAA/S scale = 3].
Bispectral index (BIS) value before and after intubation | at the time points that propofol target effect site concentration reach to 0, 2, 4, 5, 6 μg/ml, and the time points before and after intubation
  Investigators measure the Bispectral index (BIS) value at time points that propofol target effect site concentration reach to 0, 2, 4, 5, 6 μg/ml, and the time points before and after intubation.
Band power (Gamma, Beta, Alpha, Theta, and Delta waves) before and after intubation | at the time points that propofol target effect site concentration reach at 0, 2, 4, 5, 6 μg/ml, and the time points before and after intubation
  Investigators calculate band power from the data file at the time points that propofol target effect site concentration reach 0, 2, 4, 5, 6 μg/ml, and the time points before and after intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Hye-Won Shin, Ph.D., Principal Investigator — Korea University Anam Hospital, Seoul, Inchon-ro 8-gil 73, Seoul, Republic of Korea
Locations (2):
- South Korea (2):
  - Korea University Anam Hospital, Seoul, Inchon-ro 8-gil 73
  - Korea University Anam Hospital, Seoul

REFERENCES:
- [Derived] Shin HW, Kim HJ, Jang YK, You HS, Huh H, Choi YJ, Choi SU, Hong JS. Monitoring of anesthetic depth and EEG band power using phase lag entropy during propofol anesthesia. BMC Anesthesiol. 2020 Feb 26;20(1):49. doi: 10.1186/s12871-020-00964-5. PMID 32102676